CLINICAL TRIAL: NCT06383611
Title: Protocol for Expanded Access to Cyclic Irrigation of Vancomycin Hydrochloride and Tobramycin Sulfate in Patients Undergoing Exchange Arthroplasty for Periprosthetic Joint Infection of the Hip or Knee
Brief Title: Expanded Access to Cyclic Irrigation in Patients Undergoing Exchange Arthroplasty
Acronym: APEX-EAP
Status: Temporarily not available | Type: Expanded Access
Sponsor: Osteal Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OTX-0303
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Prosthetic-joint Infection
Keywords: Hip; Knee; Biofilm; Minimum biofilm eradication concentration

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Combination Product: VT-X7 Treatment System — Local antibiotic irrigation via the VT-X7 Treatment System adjuvant to two-stage exchange arthroplasty per standard of care.

SUMMARY:
The objective of the protocol is to provide access to the VT-X7 (Vancomycin, Tobramycin Exchanged in 7 Days) system for subjects with periprosthetic joint infection (PJI) of the hip or knee who lack therapeutic treatment alternatives.

ELIGIBILITY:
Inclusion Criteria:

1. Planned removal of hip or knee prosthesis as part of an exchange arthroplasty, due to hip or knee PJI. The prosthesis removed may be either i) a permanent implant or, ii) a temporary spacer implanted during a resection arthroplasty.
2. Patients who have failed a prior exchange arthroplasty.
3. Signed informed consent.
4. 22 to 84 years of age (inclusive).
5. Medical clearance for surgery.
6. Pre-enrollment diagnosis of PJI of the hip or knee per the International Consensus Meeting of Musculoskeletal Infection (ICMMI) 2018 definition of Periprosthetic Hip and Knee Infection.

Exclusion Criteria:

1. Patients who are judged by the Study Site PI to be unsuitable for the study (i.e., current medical condition that would interfere with study conduct or results or unreliable for required study follow-up).
2. Patients with bacteremia or positive bacterial blood culture in the last 30 days.
3. Patients with concurrent PJI of more than one joint.
4. Patients with ongoing active infection of an intravenous (IV) site.
5. Patients who require long-term anticoagulation or antiplatelet therapy, and for whom bridging or withholding therapy is not recommended based on the individual's clinical condition.
6. Patients with advanced renal insufficiency (i.e., chronic kidney disease (CKD) Stage 4 or 5 or patients with an estimated glomerular filtration rate (eGFR) <30 mL/min) measured within 180 days of consent.
7. Patients on chemotherapy for malignant disease.
8. Patients on systemic glucocorticoid therapy (prednisone >10 mg/day or equivalent).
9. Patients who are immunodeficient (e.g., splenectomy, sickle cell anemia, Stage 3 human immunodeficiency virus (HIV) infection, primary immunodeficiency disease), except patients who are immunodeficient due to immunosuppressive therapy.
10. Patients who have an allergy to vancomycin hydrochloride or tobramycin sulfate (Note: prior history of red man syndrome is not considered an allergy).
11. Patients who have an allergy to titanium, titanium alloys, polymethylmethacrylate or polyurethane.
12. Patients who are pregnant or planning to become pregnant in the next 30 days.
13. Patients with a fungal PJI as determined by one or more positive fluid and/or tissue cultures.
14. Patients who have a skeletal defect greater than 150 mm in length in the tibia or femur of the infected joint.
15. Patients who have a planned surgical procedure within 30 days of enrollment that can impact the conduct of the study.
16. Patients who are breastfeeding.
17. Patients who are incarcerated or are facing impending incarceration.
18. Patients who have been in treatment for substance abuse within the past year or referred to treatment for substance abuse within the past year.
19. Patients who will participate in another clinical study of an investigational drug or investigational device or have participated in another clinical study of an investigational drug or investigational device within the past 30 days that would interfere with the study results or the conduct of the study.
20. Patients receiving immunosuppressive drug therapy for bone marrow or another transplant.
21. Patients who receive therapy including any of the following biologic agents, which will not be withheld for a period beginning at least one dosing cycle (minimum 7 days) prior to planned surgery and ending at least 14 days following planned surgery:

Adalimumab (Humira) Tocilizumab (Actemra) Etanercept (Enbrel) Anakinra (Kineret) Golimumab (Simponi) Secukinumab (Cosentyx) Infliximab (Remicade) Ustekinumab (Stelara) Abatacept (Orencia) Tofacitinib (Xeljanz) Belimumab (Benlysta)

Ages: 22 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Iowa, North Liberty, Iowa
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma